CLINICAL TRIAL: NCT01692262
Title: A Phase Ib Multicentre Study of AZD5363 Monotherapy to Assess Anti-Tumour Activity,Safety,Tolerability,and Pharmacokinetics in Patients With Metastatic Castrate-Resistant Prostate Cancer (mCRPC)(PYRUS)
Brief Title: Investigating Safety, Tolerability and Efficacy of AZD5363 in Prostate Cancer.
Acronym: PYRUS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: D3610C00003; GU86
Record Dates: First submitted 2012-09-19; First posted 2012-09-25 (Estimated); Last update posted 2014-06-19 (Estimated); Status verified 2014-06

CONDITIONS: Metastatic Castrate-Resistant Prostate Cancer (mCRPC),; Efficacy,; Safety and Tolerability,; Pharmacokinetics,; Pharmacodynamics,; Tumour Response.
Keywords: Metastatic Castrate-Resistant Prostate Cancer (mCRPC),; adenocarcinoma of the prostate,; prostate cancer,; progressive disease,; advanced disease.
MeSH Terms: conditions — Prostatic Neoplasms; Disease Progression

ARMS (3):
- Part A Group 1 Intermittent (Experimental): Recruitment suspended and will not be re-opened. See intervention description below.
  Interventions: Drug: Intermittent dosing of AZD5363
- Part A Group 2 Intermittent (Experimental): Recruitment complete. See intervention description below.
  Interventions: Drug: Intermittent dosing of AZD5363
- Part B (Experimental): This part of the study will not be conducted following a review of data from Part A. See intervention description below.
  Interventions: Drug: Intermittent dosing of AZD5363

INTERVENTIONS:
Drug: Intermittent dosing of AZD5363 — Intermittent dosing of AZD5363: oral solid formulation, twice daily (480 mg bid 4 days on and 3 days off). Recruitment suspended and will not be re-opened.
  Arms: Part A Group 1 Intermittent
Drug: Intermittent dosing of AZD5363 — Intermittent dosing of AZD5363: oral solid formulation, twice daily (480 mg bid 4 days on and 3 days off). Treatment to begin on Day 1 and to continue to study withdrawal. Recruitment complete.
  Arms: Part A Group 2 Intermittent
Drug: Intermittent dosing of AZD5363 — Intermittent dosing of AZD5363: oral solid formulation, twice daily (480 mg bid 4 days on and 3 days off). Treatment to begin on Day 1 and to continue until study drug withdrawal. This part of the study will not be conducted.
  Arms: Part B

SUMMARY:
To investigate the safety, tolerability and anti-tumour activity of AZD5363, as monotherapy, in patients with metastatic Castrate-Resistant Prostate Cancer. AZD5363 will be investigated in patients who have progressed after chemotherapy (Part A) and in patients who have progressed before receiving chemotherapy (Part B).

Recruitment into Part A, Group 1 has been suspended. A new design for this group is currently being evaluated. Part A, group 2 patients (progressed after 1 or more 2nd generational anti-hormonal therapies) will receive AZD5363 480mg bid intermittently (4 days on/3days off).

Part B will only start if there is evidence of anti-tumour activity along with AZD5363 having an acceptable safety profile in Part A. Part B will be conducted in pre-chemotherapy patients on a dose and schedule selected from Part A.

DETAILED DESCRIPTION:
A Phase Ib Multicentre Study of AZD5363 Monotherapy to Assess Anti-Tumour Activity, Safety, Tolerability, and Pharmacokinetics in Patients With Metastatic Castrate-Resistant Prostate Cancer (mCRPC) (PYRUS)

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent
* Males aged 18 years and older
* Histologically confirmed adenocarcinoma of the prostate without neuroendocrine differentiation or small cell features for which no standard therapy is currently considered appropriate
* Documented evidence of Metastatic Castrate-Resistant Prostate Cancer (mCRPC)
* Part A: Patients must have received prior docetaxel-based chemotherapy for mCRPC and have a Circulating Tumour Cell score of 5;
* Part B: Patients must have progressed before receiving any chemotherapy for mCRPC;

Exclusion Criteria:

* Any prior exposure to agents which inhibit AKT as the primary pharmacological activity
* Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension, active bleeding diatheses, or active infection including hepatitis B, hepatitis C, and human immunodeficiency virus
* Spinal cord compression or brain metastases unless asymptomatic, treated, and stable and not requiring steroids
* Clinically significant abnormalities of glucose metabolism
* Major surgery within the previous 4 weeks

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2012-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Parts A and B: Anti-tumour activity by measurement of changes in circulating prostate-specific antigen (PSA) | PSA measured from baseline for every 4 weeks. Primary assessment is at 12 weeks
Parts A and B: Anti-tumour activity by measurement of changes in circulating tumour cells (CTC) | CTC measured from baseline for every 4 weeks to week 12 (primary assessment) then measured every 12 weeks
Parts A and B: Anti-tumour activity by measurement of malignant soft tissue response rate | Tumour assessments by RECIST v1.1 every 12 weeks from baseline up to disease progression or withdrawal of consent
Parts A and B: Anti-tumour activity by measurement of metastatic bone disease status | Bone lesion assessments by bone scan (PCWG2) criteria every 12 weeks from baseline up to disease progression or withdrawal of consent.

SECONDARY OUTCOMES:
Parts A and B: Safety and tolerability of AZD5363 in terms of adverse events, serious adverse events (including death) and safety measures: ECG, ECHO/MUGA, physical examination, pulse, blood pressure, weight and laboratory variables | Routine safety assessments, throughout the period that patients receive AZD5363 up to 28 days following discontinuation of study treatment.
Parts A and B: AZD5363 PK: time to maximum plasma concentration, terminal rate constant,terminal half life, area under plasma concentration time curve, plasma clearance & volume of distribution | Multiple AZD5363 PK blood sample assessments.AZD5363 plasma concentration blood samples will be taken on Day 1(pre-dose,2,4,8 hours post-dose);D2(pre-dose);D8(continous) or D11(intermittent) (pre-dose and at 2,4,and 8 hours post-dose);D15,Cyc
Parts A and B: Plasma concentrations of pharmacodynamic (PD) biomarker | Multiple PD blood sample assessments.PD blood samples will be taken on the same schedule as PK sample and then Day 1 of every 12 weeks thereafter, and at the discontinuation visit
Parts A and B: Progression-free survival (PFS) | Tumour assessments by RECIST v1.1 every 12 weeks from baseline up to disease progression or withdrawal of consent.
Parts A and B: Quality of life (QoL) | QOL will be documented from date of randomization and for 12 weeks.
  EORTC QLQ-C15-PAL, EORTC QLQ-PR25, and EORTC QLQ-BM22 Questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Paul Stockman, MBCHB, PHD, Study Director — AstraZeneca
Locations (8):
- United States (5):
  - Research Site, Sarasota, Florida
  - Research Site, Boston, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Hackensack, New Jersey
  - Research Site, Nashville, Tennessee
- United Kingdom (3):
  - Research Site, Cardiff, Wales
  - Research Site, London
  - Research Site, Southampton